CLINICAL TRIAL: NCT02050100
Title: Biomarkers for Diagnosis of Lung Cancer
Status: Completed | Type: Observational
Sponsor: SK Medical (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SKTCTCH0001
Record Dates: First submitted 2014-01-20; First posted 2014-01-30 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer; Lung Neoplasm
Keywords: primary lung adenocarcinoma Stages I, II, IIIA, IIIB; squamous cell carcinoma Stages I, II, IIIA, IIIB; benign non-calcified pulmonary nodules; early detection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two 10ml blood samples (serum and plasma) from the patient will be analyzed for protein biomarkers associated with lung cancer diagnosis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung Cancer: Early-late stage primary lung cancer
- Lung Neoplasm: Benign non-calcified pulmonary nodules

SUMMARY:
The study goal is to collect blood samples from individuals at risk for lung cancer in order to identify protein markers for diagnosis of lung cancer in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Patients referred to pulmonologists, oncologists, or thoracic surgeons for diagnosis of suspicious pulmonary nodules as either lung cancer or benign and undergoing bronchoscopic biopsy
* Patients will be enrolled if the result of the bronchoscopic biopsy is a diagnosis of NSCLC or benign pulmonary nodule
* Cases: Patients with untreated non-small cell lung cancer, i.e. primary lung adenocarcinoma or squamous cell carcinoma of early
* Computed tomography or X-Ray is available and shows a suspicious pulmonary nodule
* A biopsy or surgical resection to clarify the nature of the lung nodule is available (NSCLC or benign, including histological diagnosis) in both groups
* Controls: Patients must be available for a 6 month follow-up to confirm benign diagnosis
* A serum and plasma sample was collected prior to any treatment of the lung nodule beyond biopsy
* No other cancer diagnosis in the last 5 years excluding non-melanoma skin cancer
* Patients must be fully informed of the investigational nature of the procedure and sign an informed consent.

Exclusion Criteria:

* Prior treatment for lung cancer by chemotherapy or surgery (excluding biopsy)
* Patients with benign nodules who are not able or willing to have a 6-month follow-up visit to confirm benign diagnosis
* Diagnosis or treatment of other cancer in the last 5 years excluding non-melanoma skin cancer. In the judgment of the clinical investigator, patients who are likely to be non compliant or uncooperative during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 patients will be recruited from hospital pulmonary clinics. The study participants will have pulmonary nodules suspicious for lung cancer and a bronchial biopsy diagnosis of NSCLC or probable benign. Approximately half of the patients will be cases and half controls.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Identification of blood biomarkers for detection of lung cancer | 6 months after enrollment
  SK Telecom will utilize 15 single-plex quantitative Polymerase Chain Reaction (qPCR) assays to analyze an initial set of 300 clinical samples in China. SomaLogic will analyze these samples on the SOMAscan array (>1000 proteins) for additional lung cancer biomarker candidates.

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue Bai, M.D, Ph.D., Principal Investigator — Zhongshan Hospital Fudan Universit; Xiaoju Zhang, M.D., Principal Investigator — Henan Provincial People's Hospital; Muyun Zhu, M.D., Principal Investigator — Northern Jiangsu People's Hospital; Kai Wang, MD, Principal Investigator — The Second Affliated Hospital of Zhejiang University School of Medicine; Zuke Xiao, MD, Principal Investigator — Jiangxi Provincial People's Hopital
Locations (5):
- China (5):
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The Second Affliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhongshan Hospital Fudan University, Shanghai
  - Henan province People's hospital, Zhengzhou